CLINICAL TRIAL: NCT05036187
Title: Using the Multiphase Optimization Strategy to Optimize a Culturally Tailored Online Behavioral Weight Loss Intervention for Sexual Minority Women: Pilot Study
Brief Title: Refining Novel Culturally Tailored Behavioral Weight Loss Treatment Components for Sexual Minority Women With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 1550062; K23MD015092 (NIH)
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: Sexual minority women; LGBTQ health; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: After a pre-piloting phase (consisting of initial content piloting, interviews, and intervention refinement; anticipated n=12), participants (anticipated n=8) will receive the online weight loss treatment and will be randomized to receive 0-3 novel intervention components (targeting minority stress, negative body image, and social support) over the 3-month period. Participants will complete quantitative and qualitative assessments of intervention acceptability and appropriateness post-treatment.
  Enrollment for both the pre-piloting phases (anticipated n=12) and open pilot trial phase (anticipated n=8) are reported here.
Masking Description: There is no masking during the pilot phase where the goal is to improve the program's acceptability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Weight Loss Program Only (Experimental): Participants complete an online behavioral weight loss program.
  Interventions: Behavioral: Behavioral Weight Loss Intervention
- Weight Loss Program + Coping with Stress Program (Experimental): Participants complete (1) an online behavioral weight loss program and (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Minority Stress Intervention
- Weight Loss Program + Coping with Stress Program + Body Image Program (Experimental): Participants complete (1) an online behavioral weight loss program, (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss, and (3) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Minority Stress Intervention; Behavioral: Negative Body Image Intervention
- Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program (Experimental): Participants complete (1) an online behavioral weight loss program, (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss, (3) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts, and (4) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Minority Stress Intervention; Behavioral: Negative Body Image Intervention; Behavioral: Social Support Intervention
- Weight Loss Program + Body Image Program + Social Support Program (Experimental): Participants complete (1) an online behavioral weight loss program, (2) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts, and (3) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Negative Body Image Intervention; Behavioral: Social Support Intervention
- Weight Loss Program + Coping with Stress Program + Social Support Program (Experimental): Participants complete a (1) online behavioral weight loss program, (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss, and (3) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Minority Stress Intervention; Behavioral: Social Support Intervention
- Weight Loss Program + Body Image Program (Experimental): Participants complete (1) an online behavioral weight loss program and (2) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Negative Body Image Intervention
- Weight Loss Program + Social Support Program (Experimental): Participants complete (1) an online behavioral weight loss program and (2) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts.
  Interventions: Behavioral: Behavioral Weight Loss Intervention; Behavioral: Social Support Intervention

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Intervention — Rx Weight Loss: PRIDE is a fully automated online behavioral obesity treatment that is tailored for sexual minority women and involves viewing 12 online video lessons delivered each week, self-monitoring body weight, calorie intake, and physical activity levels, and receiving personalized automated weekly feedback on progress toward goals.
Behavioral: Minority Stress Intervention — The Minority Stress Intervention is designed to help sexual minority women cope with stress and stigma (e.g., due to weight, sexual orientation, gender). In this program, participants watch online video lessons that teach cognitive and behavioral strategies for coping with minority stress so that it may have less of an influence on participants' weight and well-being.
  Other Names: Coping with Stress Program
  Arms: Weight Loss Program + Coping with Stress Program; Weight Loss Program + Coping with Stress Program + Body Image Program; Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Social Support Program
Behavioral: Negative Body Image Intervention — The Negative Body Image Intervention is designed to help participants improve their body image. In this program, participants will watch online video lessons that provide education on queer women's body image and teach cognitive and behavioral strategies for improving your body image (regardless of your weight) to reduce its influence on your health.
  Other Names: Body Image Program
  Arms: Weight Loss Program + Body Image Program; Weight Loss Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Body Image Program; Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program
Behavioral: Social Support Intervention — The Social Support Intervention provides online opportunities for participants to receive more social support as they work toward their weight loss goals. Participants receive education on the importance of social support for weight management, they can earn badges for completing program milestones, and they gain access to a private online forum to get support and advice from other participants.
  Arms: Weight Loss Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Social Support Program; Weight Loss Program + Social Support Program

SUMMARY:
Obesity disproportionately impacts sexual minority women. Behavioral weight loss programs are the gold standard treatment for mild to moderate obesity. The investigators have developed an online behavioral weight loss program that is effective, low-cost, and highly scalable. However, existing research suggests that tailoring treatment to address 3 well-established weight loss barriers in sexual minority women will be critical for maximizing the relevance and efficacy of behavioral weight loss for this group. The goal of the first phase of this K23 is to develop 3 novel treatment components targeting sexual minority women's weight loss barriers (i.e., minority stress, low social support, and negative body image), to pilot the program in sexual minority women with overweight/obesity, and to conduct individual qualitative interviews to elicit feedback on the intervention's acceptability, cultural relevance, usability, and feasibility that will be used to refine the program. After a pre-piloting phase (consisting of initial content piloting, interviews, and intervention refinement; anticipated n=12), 8 participants will pilot the full 3-month weight loss program and will be randomized to pilot 0-3 novel tailored components (targeting minority stress, negative body image, and social support) over the 3-month period. Participants will complete quantitative and qualitative assessments of intervention acceptability and appropriateness post-treatment and the intervention will be refined.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth and currently identify as female
* Self-identify a minority sexual orientation (e.g.,lesbian, bisexual)
* BMI>25kg/m2
* 18-70 years old
* Interested in losing weight
* Regular internet and e-mail access
* Fluent in English

Exclusion Criteria:

* Significant weight loss within past 6 months (>5%)
* Unable to participate in moderate physical activity
* Currently enrolled in a weight loss program
* Currently taking weight-loss medication
* Currently pregnant or trying to get pregnant
* Participated in a previous Phase of this study
* Reports a serious mental/physical health condition that would increase potential risks of treatment to the participant (e.g., active symptoms of psychosis, suicidality, mania, alcohol/substance use, or a medical condition that is serious, active, unstable, and degenerative (e.g., CHF)).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who currently self-identify as female are being recruited.
Enrollment: 28 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability | Week 12 (post-treatment)
  A measure of intervention acceptability adapted from the Acceptability of Intervention (AIM) measure will assess acceptability outcomes post-treatment. Qualitative data on intervention acceptability and cultural appropriateness will also be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared as follows:
  * Results will be submitted to ClinicalTrials.gov within appropriate timelines.
  * Quantitative data will be published in peer-reviewed manuscripts that will be submitted to PubMed Central upon acceptance.
  * Study results will be presented to the scientific community at national conferences relevant to obesity and sexual minority health.
  * Aggregate quantitative data may be requested from other researchers 5 years after the completion of the primary endpoint by contacting Dr. Panza. If there are no restrictions imposed by institutional policies, local IRBs, or laws/regulations, the investigators will make de-identified data available to a requester within the context of a clear data-sharing agreement Qualitative data will not be shared other than de-identified qualitative data that is published as part of peer-reviewed manuscripts.

DOCUMENTS (1):
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT05036187/ICF_000.pdf